CLINICAL TRIAL: NCT00631540
Title: REFORM Clinical Study: Treatment of Renal Artery Stenosis With the Formula Balloon-Expandable Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-581; FRUS
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2011-05-19 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-11

CONDITIONS: Renal Artery Stenosis
Keywords: renal artery stenosis; hypertension; renovascular; renal artery blockage; renal artery disease; renal arteries; angioplasty renal artery; renal artery stent; renal artery doppler; renovascular hypertension; kidney stenosis; renal artery; stent; stenting; kidney disease; renal failure; atherosclerosis; arterial hypertension; stenosis
MeSH Terms: conditions — Renal Artery Obstruction; Hypertension; Hypertension, Renovascular; Kidney Diseases; Renal Insufficiency; Atherosclerosis; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): renal artery stenting
  Interventions: Device: Formula Balloon-Expandable Stent

INTERVENTIONS:
Device: Formula Balloon-Expandable Stent — renal artery stenting
  Other Names: renal artery revascularization

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of the Formula Balloon-Expandable Stent in treatment of renal artery stenosis.

ELIGIBILITY:
Key Inclusion Criteria:

* renal artery stenosis
* appropriate size and location of the lesion
* suboptimal angioplasty

Key Exclusion Criteria:

* less than 18 years old
* failure or inability to give informed consent
* simultaneously participating in another drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-02; Primary Completion 2010-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bersin, MD, Principal Investigator — Swedish Medical Center
Locations (7):
- United States (7):
  - Munroe Regional Medical Center, Ocala, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Lenox Hill Hospital, New York, New York
  - Wake Med Raleigh Campus, Raleigh, North Carolina
  - Fairfield Medical Center, Lancaster, Ohio
  - Pinnacle Health at Harrisburg, Harrisburg, Pennsylvania
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Bersin RM, Ansel G, Rizzo A, Bob Smouse H, Sinha S, Sachar R, Dave R, Weinstock BS, Feldman R, Roubin GS. Nine-month results of the REFORM study: a prospective, single-arm, multicenter clinical study of the safety and effectiveness of the Formula balloon-expandable stent for treatment of renal artery stenosis. Catheter Cardiovasc Interv. 2013 Aug 1;82(2):266-73. doi: 10.1002/ccd.24481. Epub 2013 Mar 25. PMID 22581488

RESULTS

PARTICIPANT FLOW:
Groups:
- Formula™ Balloon-Expandable Renal Stent: renal artery stenting
Period: Overall Study
Arm/Group | Formula™ Balloon-Expandable Renal Stent
Started | 100
Completed | 86
Not Completed | 14
Not completed — Withdrawal by Subject | 5
Not completed — Death | 4
Not completed — Lost to Follow-up | 2
Not completed — Core Lab Data Unavailable | 3

BASELINE CHARACTERISTICS:
Arm/Group | Formula™ Balloon-Expandable Renal Stent
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 44
Region of Enrollment [Number; unit: Participants]
  United States | 100
Hypertension [Number; unit: Participants] — Pre-hypertension: Systolic 120-139 mmHg, Diastolic 80-89 mmHg Stage 1: Systolic 140-159 mmHg, Diastolic 90-99 mmHg Stage 2: Systolic >160 mmHg, Diastolic > 100 mmHg If systolic and diastolic pressures were in different categories, the higher category was chosen.
  Participants
    Hypertension | 97
    No Hypertension | 3
Renal Insufficiency [Number; unit: Participants] — Renal Insufficiency was defined by the physician, based on the patient's medical history.
  Participants
    Renal Insufficiency | 46
    No Renal Insufficiency | 54
Congestive Heart Failure [Number; unit: Participants]
  Congestive Heart Failure | 26
  No Congestive Heart Failure | 74
Serum Creatinine [Mean (Standard Deviation); unit: mg/dl] | 1.3 (0.5)
Estimated Glomerular Filtration Rate [Mean (Standard Deviation); unit: ml/min] | 60.7 (28.8)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 150.3 (20.6)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 73.9 (12.9)
Number of Antihypertensive Medications per Patient [Mean (Standard Deviation); unit: Antihypertensive Medications] | 2.7 (1.2)
Percent Stenosis at Baseline [Mean (Standard Deviation); unit: Percent] — Baseline stenosis was determined by angiography.
  Percent
    Core Lab | 57.4 (13.8)
    Site Reported | 82.5 (8.1)

OUTCOME MEASURES:

1. Primary Outcome: Primary Patency of the Treated Renal Artery
Description: Based on ultrasound images assessed by core lab.
Time Frame: 9 Months
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Formula™ Balloon-Expandable Renal Stent
Number analyzed (Participants) | 86
Number analyzed (Lesions) | 99
Lesions | 91
Statistical Analysis 1: Comparison: Formula™ Balloon-Expandable Renal Stent; Alternative hypothesis is 9-month primary patency rate greater than 60%; Test type: Superiority or Other; p < 0.0001, Z-test, 1-sided; Mean Patency Rate = 91.7, 95% CI 2-sided [84.2 to 95.9] — GEE model estimate

2. Secondary Outcome: Number of Participants With 30-day Major Adverse Events
Description: Clinical Events Committee Adjudicated Death, Clinical Events Committee Adjudicated Q-wave MI, Clinically-driven Target Lesion Revascularization, Clinical Events Committee Adjudicated Significant Embolic Events.
Time Frame: 30 Days
Population: 1 participant withdrew and 1 participant was lost to follow-up prior to 30 days.
Measure: Number; unit: Participants
Arm/Group | Formula™ Balloon-Expandable Renal Stent
Number analyzed (Participants) | 98
Participants | 0

3. Secondary Outcome: Number of Participants With 9-month Major Adverse Events
Description: as for outcome 2
Time Frame: 9 Months
Population: 3 participants withdrew, 4 died, and 1 was lost to follow-up prior to 300 days.
Measure: Number; unit: Participants
Arm/Group | Formula™ Balloon-Expandable Renal Stent
Number analyzed (Participants) | 92
Participants
  Clinically-driven Target Lesion Revascularization | 2
  Clinical Events Committee (CEC) Adjudicated Death | 0
  CEC Adjudicated Significant Embolic Events | 0
  Clinical Events Committee Adjudicated Q-wave MI | 0

4. Secondary Outcome: Technical Success
Description: Successful delivery and deployment of a Formula™ Balloon-Expandable Stent at index procedure.
Time Frame: Prior to Discharge
Measure: Number; unit: Percentage of Participants
Arm/Group | Formula™ Balloon-Expandable Renal Stent
Number analyzed (Participants) | 100
Percentage of Participants | 97

5. Secondary Outcome: Acute Procedural Success
Description: < 30% residual stenosis post-procedure by core lab analysis and no Major Adverse Events before discharge.
Time Frame: Prior to Discharge
Population: 1 participant did not have core lab assessment for stenosis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Formula™ Balloon-Expandable Renal Stent
Number analyzed (Participants) | 99
Percentage of Participants | 95

6. Secondary Outcome: 30-day Clinical Success
Description: < 30% residual stenosis post-procedure by core lab analysis and no Major Adverse Events within 30 days.
Time Frame: 30 Days
Population: 1 participant was lost to follow-up, 1 participant withdrew, 1 participant did not have core lab assessment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Formula™ Balloon-Expandable Renal Stent
Number analyzed (Participants) | 97
Percentage of Participants | 95

ADVERSE EVENTS:
Arm/Group | Formula™ Balloon-Expandable Renal Stent
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 11/99
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Formula™ Balloon-Expandable Renal Stent (N=99)
Arrhythmias (30 days to 9 months) (Cardiac disorders) | 6 (7) — 1 participant withdrew, 1 participant was lost to follow-up who experienced adverse events but were not reported here due to < 5%
Cardiac Ischemia (30 days to 9 months) (Cardiac disorders) | 6 (6) — 1 participant withdrew, 1 participant was lost to follow-up who experienced adverse events but was not reported here due to < 5%

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days